CLINICAL TRIAL: NCT05855512
Title: Impact of Nurse-led Intervention on Asthma Control in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12/2017/12
Record Dates: First submitted 2023-02-03; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2020-08

CONDITIONS: Asthma in Children

STUDY DESIGN:
Intervention Model Description: Intervention and control group
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled group (No Intervention): No intervention was given, only the material was provided in the form of a booklet
- Interventional Group (Experimental): The nursing educational intervention sessions were conducted, and the material was provided in the form of a booklet
  Interventions: Other: Nursing Educational Intervention

INTERVENTIONS:
Other: Nursing Educational Intervention — Nursing Educational Intervention
  Arms: Interventional Group

SUMMARY:
This randomized control trial design (RCT) study was conducted on children aged 6 -11 years

DETAILED DESCRIPTION:
This randomized control trial design study was conducted on children aged 6 -11 years, visiting the pediatric outpatient department and emergency at Dr. Ruth Pfau Civil Hospital Karachi.

For the experimental group, a nursing educational intervention session was conducted with the patient and family/caregiver by the principal investigator, and a doctor provided the usual care/treatment. In contrast, the control group received only the usual care/treatment provided by the doctor.

For the control group, educational material on asthma was provided in a booklet according to Global Initiative of Asthma (GINA) guidelines. Pre Childhood-Asthma Control Test (C-ACT) score of participants was measured before the intervention, and post-C-ACT score measurement was made after one month using the same questionnaires and C-ACT tool.

ELIGIBILITY:
Inclusion Criteria:

* Children between the aged 6 to 11 years
* Have asthma diagnosed by a physician at least 6-month back
* Uncontrolled asthma based on C-ACT score 19 or less 19.

Exclusion Criteria:

* Chronic respiratory illnesses like T.B. cystitis and fibrosis.
* Sinusitis,
* Gastrointestinal reflux disease,
* Rhinitis

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Childhood asthma control test (C-ACT) Score | 4 weeks
  C-ACT Score was measured in both controlled and intervention groups and compared the difference between pre-intervention and post-intervention
Number of times got Admissions due to asthma in the last 4 weeks | 4 weeks
  Using the same questionnaire number of admissions was compared to the difference between pre-intervention and post-intervention by the mean and standard deviation

SECONDARY OUTCOMES:
Number of times visited emergency due to asthma in last 4 weeks | 4 weeks
  Using the same questionnaire number of admissions was compared to the difference between pre-intervention and post-intervention by the mean and standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Waqas Farooqi, PhD, Study Director — Dow University of Health Sciences Karachi
Locations (1):
- Civil Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No